CLINICAL TRIAL: NCT04120454
Title: An Investigator-Sponsored Phase 2 Single Arm Trial of Ramucirumab and Pembrolizumab in Patients With EGFR Mutant Non-Small Cell Lung Cancer
Brief Title: Ramucirumab and Pembrolizumab for the Treatment of EGFR Mutant Recurrent or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Asrar Alahmadi, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19132; NCI-2019-05348 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ramucirumab, pembrolizumab) (Experimental): Patients receive ramucirumab IV over 60 minutes and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Biological: Ramucirumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Ramucirumab — Given IV
  Other Names: anti-VEGFR-2 fully human monoclonal antibody IMC-1121B; Cyramza; IMC-1121B; LY3009806; Monoclonal Antibody HGS-ETR2

SUMMARY:
This phase II trial studies how well ramucirumab and pembrolizumab work in treating EGFR mutant non-small cell lung cancer that has come back (recurrent) or spread to other places in the body (metastatic) while on systemic therapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ramucirumab, a drug which has anti-angiogenic and pleotropic immunomodulatory effects and may synergize with the effect of an anti-PD-1 agent. The study investigates the effect of targeted anti-antitumor activity of immune checkpoint inhibitor pembrolizumab and immune-suppressive activity of VEGF-inhibitor ramicirumab to evaluate the efficacy and the tolerability of the combination.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate response rate of the combination of ramucirumab and pembrolizumab in EGFR mutant non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVE:

I. To evaluate safety, tolerability, and survival for patients receiving pembrolizumab and ramucirumab.

EXPLORATORY OBJECTIVE:

I. To characterize predictive immunologic biomarkers of response in tissue and peripheral blood of patients receiving ramucirumab and pembrolizumab combination therapy.

OUTLINE:

Patients receive ramucirumab intravenously (IV) over 60 minutes and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥18 years
2. Histologically confirmed recurrent or metastatic non-small cell carcinoma of the lung with sensitizing EGFR mutations. Exon 20 resistance mutations will not be permitted but uncommon sensitizing mutations are allowed.
3. Prior Systemic Anticancer Therapy: Neo/adjuvant therapy or prior therapy for locally advanced disease will be permitted. Patients with prior exposure to PD/PD-L1 inhibitors will be excluded. No limit on prior EGFR TKIs (erlotinib, gefitinib, afatinib, dacomitinib or osimertinib). Prior chemotherapy for metastatic disease is permitted only. A 7 day washout period or four half-lives after the last treatment dose, whichever is longer, is required for TKI. A 4 week washout is required for cytotoxic chemotherapy.
4. Measurable disease per RECIST criteria
5. ECOG performance status of 0-1
6. Adequate organ function, hematologic, hepatic, renal and coagulation parameters as defined in the protocol.
7. Because the teratogenicity of ramucirumab is not known, the patient, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods).
8. Female patients of childbearing potential must have a negative serum pregnancy test within 72 hours prior to first dose of protocol therapy.

Exclusion Criteria

1. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
2. Known active chronic infections - HIV/AIDS, known active Hepatitis B or C. Known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
3. Cirrhosis (Child-Pugh B or worse) or cirrhosis with history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis.
4. Prior exposure to ramucirumab.
5. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
6. Any Grade 3-4 GI bleeding within 3 months prior to first dose of protocol therapy.
7. History of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy.
8. Patients receiving dipyridamole, clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
9. Uncontrolled CNS metastases. Patients with treated brain metastases are eligible if they were clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) ending at least 2 weeks prior to first dose of study treatment, or after surgical resection performed at least 28 days prior to first dose of study treatment. The patient must have no evidence of Grade ≥1 CNS hemorrhage based on pretreatment MRI or IV contrast CT scan (performed within 28 days before first dose of study treatment). Note: Patients who received systemic therapy that adequately and appropriately treated CNS metastases, including tyrosine kinase inhibitors, are eligible provided that CNS disease control is confirmed by pretreatment MRI within 28 days of receiving first dose of study treatment.
10. Hemoptysis (defined as bright red blood or ≥ 1/2 teaspoon) within 2 months prior to first dose of protocol therapy or with radiographic evidence of intratumor cavitation or has radiologically documented evidence of major blood vessel invasion or encasement by cancer.
11. Uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
12. Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy.
13. Major surgery within 28 days or device placement within 7 days prior to the first dose of protocol therapy. Patient has elective or planned major surgery to be performed during the course of the clinical trial.
14. Serious or non-healing wound, ulcer, or bone fracture within 28 days of study treatment.
15. Prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation.
16. Small cell or mixed (small cell/non-small cell) lung cancer
17. Pregnancy or breastfeeding.
18. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
19. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
20. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
23. Active infection requiring systemic therapy.
24. Known history of active TB (Bacillus Tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asrar Alahmadi, MBBS, MAS-CR, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response rate will be evaluated with computed tomography (CT) scans every 2 cycles and tumor measurements using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Immune RECIST (iRECIST) will also be assessed.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
Number analyzed (Participants) | 6
percentage of participants | 0

2. Secondary Outcome: Number of Adverse Events
Description: Common Terminology Criteria for Adverse Events version 4.0 will be used for adverse event grading. Attributions of causality will be assessed by the primary treating physician. Frequency and severity of adverse events and tolerability of the regimen will be collected and summarized by descriptive statistics for each of the disease cohorts.
Time Frame: Up to 2 years
Measure: Number; unit: Number of Events
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
Number analyzed (Participants) | 6
Number of Events
  Lymphocyte count decreased | 4
  Activated partial thromboplastin time prolonged | 4
  Alanine aminotransferase increased | 3
  Alkaline phosphatase increased | 2
  Anemia | 3
  Anorexia | 2
  Arthralgia | 1
  Aspartate aminotransferase increased | 4
  Cognitive impairment | 1
  Constipation | 2
  Diarrhea | 1
  Dysgeusia | 3
  Dysphagia | 1
  Dyspnea | 2
  Edema limbs | 3
  Encephalopathy | 2
  Epistaxis | 1
  Fall | 1
  Fatigue | 7
  Generalized muscle weakness | 1
  Headache | 2
  Hematuria | 2
  Hypercalcemia | 1
  Hyperglycemia | 3
  Hypernatremia | 1
  Hypertension | 4
  Hyperthyroidism | 1
  Hypoalbuminemia | 5
  Hypocalcemia | 1
  Hypokalemia | 1
  Hyponatremia | 9
  Hypoxia | 1
  Imbalance | 1
  Infusion related reaction | 1
  INR increased | 4
  Bacteriuria | 1
  Localized Edema | 1
  Mucositis | 1
  Myalgia | 1
  Nausea | 1
  Neuralgia | 2
  Osteoporosis | 1
  Pericardial effusion | 1
  Pleural effusion | 1
  Pneumothorax | 1
  Productive cough | 2
  Proteinuria | 2
  Thromboembolic event | 1
  Rash maculo-papular | 2
  Nephrotic syndrome | 1
  Hemoptysis | 2
  Sinus tachycardia | 1
  Urinary incontinence | 1
  Vomiting | 3
  Weight gain | 3
  Weight loss | 2
  Confusion | 1

3. Secondary Outcome: Clinical Benefit Rate (Complete Response + Partial Response + Stable Disease)
Description: Clinical benefit rate will be evaluated with CT scans every 2 cycles and tumor measurements using RECIST 1.1 criteria. iRECIST will also be assessed.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
Number analyzed (Participants) | 6
percentage of participants | 50

4. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier curves will be calculated to estimate progression-free survival.
Time Frame: From the date of study registration to the date of progressive disease, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
Number analyzed (Participants) | 6
months | 1.4 [1.13 to NA] — There was insufficient data to determine the upper limit

5. Secondary Outcome: Overall Survival
Description: Kaplan-Meier curves will be calculated to estimate overall survival.
Time Frame: From the date of study registration to the date of death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
Number analyzed (Participants) | 6
months | 7.03 [5.57 to NA] — There was insufficient data to determine the upper limit

6. Other Pre Specified Outcome: Tumor Immunoprofile
Description: Measured by immunohistochemistry, including tumor infiltrating lymphocytes and T cell receptor (TCR) immunosequencing (immunoSEQ) and relationship to clinical outcomes, including response rate. TCR immunoSEQ data will be summarized for each patient for T-cell clonality difference, descriptive statistics and confidence interval will be obtained across patients.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Circulating Immune Cell Profiles in Response to Treatment and in Relation to Clinical Response
Description: Measured using 10-color 65 marker multiplex Clinical Laboratory Improvement Act-certified IMMUNOME flow cytometry profile on peripheral blood samples. For immune cell subpopulation data by flow cytometry, will identify differences between the paired peripheral blood mononuclear cell samples from the same patients.
Time Frame: Up to 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Circulating VEGF Levels
Description: Will evaluate correlation with clinical response. A bivariate plot will be used to describe the relationship between response rate and peak VEGF via enzyme-linked immunosorbent assay over time.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 2 years
Arm/Group | Treatment (Ramucirumab, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ramucirumab, Pembrolizumab) (N=6)
Aspartate aminotransferase increase (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ramucirumab, Pembrolizumab) (N=6)
Lymphocyte count decreased (Investigations) | 4 (4)
Activated partial thromboplastin time (Investigations) | 1 (4)
Alanine aminotransferase increased (Investigations) | 1 (3)
Alkaline phosphatase increased (Investigations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 4 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Imbalance (General disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
INR (International Normalized Ratio of prothrombin time) Increased (Investigations) | 2 (4)
Bacteriuria (Investigations) | 1 (1)
Localized edema (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Weight gain (Investigations) | 1 (3)
Weight loss (Investigations) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04120454/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04120454/ICF_001.pdf